CLINICAL TRIAL: NCT04573777
Title: Reducing Intracranial atheroSclErosis With Repatha
Acronym: RISER
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Funding Discontinued
Sponsor: University of California, Los Angeles (Other)
Collaborators: Amgen (Industry)
Responsible Party: Principal Investigator, David Liebeskind, Principal Investigator, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00121763; NCT04573010 (obsolete NCT alias)
Record Dates: First submitted 2020-09-28; First posted 2020-10-05 (Actual); Results first posted 2023-03-15 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-02

CONDITIONS: Ischemic Stroke
Keywords: Intracranial Atherosclerosis
MeSH Terms: conditions — Ischemic Stroke; Intracranial Arteriosclerosis | interventions — evolocumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Intervention Repatha (Experimental)
  Interventions: Drug: Repatha

INTERVENTIONS:
Drug: Repatha — 140 MG in 1 ML Prefilled Syringe PCSK9 Inhibitor

SUMMARY:
The purpose of this study will be to understand the underlying mechanism by which PCSK9 inhibition reduces the rate of ischemic stroke seen in the pivotal studies that led to its FDA approval for ASCVD such as ischemic stroke. Those trials (FOURIER and ODYSSEY) enrolled almost 50,000 patients and showed that PCSK9 inhibition therapy is safe and effective. The investigators hypothesize that PCSK9 inhibition lowers the rate of stroke by reducing atherosclerotic plaque, which would be particularly beneficial for patients with intracranial atherosclerosis, who have the highest rate of recurrent stroke of any stroke mechanism.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, ≥ 18 years of age
* History of ischemic stroke, defined as an episode of neurological dysfunction caused by focal cerebral, spinal, or retinal infarction (American Heart Association definition).
* Large vessel atherosclerosis of an intracranial artery in the circle of Willis with 50-99% stenosis by WASID criteria (percent stenosis = (1-[diameter stenosis/diameter normal]) x 100%) on MRA, CTA or DSA

  ------ Eligible arteries: vertebral (V4), basilar, PCA (P1, P2), MCA (M1, M2), tICA, ACA (A1)
* Current statin use or contraindication to statin
* Fasting LDL-C ≥ 70 mg/dL or LDL-C ≥ 60 mg/dL if lipoprotein (a) > 30 mg/ dL

Exclusion Criteria:

Gadolinium or PCSK9 inhibitor allergy

* Acute or chronic kidney disease with eGFR<30 ml/min/1.73m2
* Pacemaker or other MRI contraindications per American College of Radiology guidelines
* Inability to return for 78 week follow-up clinic visit and vwMRI

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-04-23 (Actual); Primary Completion 2021-12-16 (Actual); Study Completion 2021-12-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- UCLA, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention Repatha
Started | 10
Completed | 0
Not Completed | 10

BASELINE CHARACTERISTICS:
Arm/Group | Intervention Repatha
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Stenosis
Description: Measured on ToF MRA, CE-MRA, T1 Dante
Time Frame: 1.5 years
Population: Outcome data were not collected due to early termination
Arm/Group | Intervention Repatha
Number analyzed (Participants) | 0

2. Secondary Outcome: Percent Atheroma Volume
Description: Measured on ToF MRA, CE-MRA, T1/T2/PD Dante
Time Frame: 1.5 years
Population: Study funding was terminated before reaching the analysis phase of the study. No participants made it to 1.5 years. Outcome data were not collected due to early termination
Arm/Group | Intervention Repatha
Number analyzed (Participants) | 0

3. Other Pre Specified Outcome: Ischemic Stroke
Description: Adjudicated
Time Frame: 1.5 years
Population: Study funding was terminated before reaching the analysis phase of the study. No participants made it to 1.5 years
Arm/Group | Intervention Repatha
Number analyzed (Participants) | 0

4. Other Pre Specified Outcome: ITA
Description: Adjudicated
Time Frame: 1.5 years
Population: Study funding was terminated before reaching the analysis phase of the study. No participants made it to 1.5 years
Arm/Group | Intervention Repatha
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 8 Months
Description: Study has concluded prematurely and we are no longer tracking adverse event for study population
Arm/Group | Intervention Repatha
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-01): https://cdn.clinicaltrials.gov/large-docs/77/NCT04573777/Prot_SAP_001.pdf